CLINICAL TRIAL: NCT07037797
Title: Phased-Array Versus Curvilinear Probe for FAST Ultrasonography
Acronym: PAC-FAST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Memorial France Etats-Unis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-2024-001; 2024-A00914-43 (Other: ID RCB)
Record Dates: First submitted 2025-05-13; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Chest Trauma; Abdominal Trauma
Keywords: chest trauma; abdominal trauma
MeSH Terms: conditions — Thoracic Injuries; Abdominal Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Curvilinear probe then phased-array probe (Experimental): The first probe used is the curvilinear following by the phased-array probe
  Interventions: Diagnostic Test: Order of the FAST echography
- Phased-array probe then curvilinear probe (Experimental): The first probe used is the phased-array probe following by the curvilinear probe
  Interventions: Diagnostic Test: Order of the FAST echography

INTERVENTIONS:
Diagnostic Test: Order of the FAST echography — Randomisation of the order in which probes are used

SUMMARY:
Background:

FAST ultrasound is a crucial technique in emergency medicine, enabling rapid assessment of trauma patients.

By allowing visualization of an effusion in a trauma patient in a far more sensitive and specific way than clinical examination, it enables informed decisions to be made on therapeutics, technical gestures, but also the potential receiving service.

Arbitrarily, FAST ultrasound is taught with the cardiac probe (phased-array) and the abdominal probe (curvilinear). The difference in use of these two probes varies according to operator and team, with no figures available.

No recent study has been conducted on the possibility of better diagnostic performance of FAST with a curvilinear versus phased-array probe.

Objective:

The main objective of this project is to evaluate and compare the diagnostic performance of FAST ultrasound using a phased-array probe versus a curvilinear probe in the detection of effusions in trauma patients (FAST protocol).

Materials and methods:

Prospective, interventional, multicenter, randomized study.

Hypothesis tested:

FAST-ultrasound with a curvilinear probe improves diagnostic performance compared with FAST-ultrasound with a phased-array probe.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients attending emergency departments in investigating centers
* Age ≥ 18 years
* Indication retained for FAST-ultrasound by the emergency physician in charge of the patient
* Patient affiliated to the French Social Security system or equivalent

Exclusion Criteria:

* Patients undergoing treatment limitation or discontinuation
* Pregnant, parturient or breast-feeding women
* Patients deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2660 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-02 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance | From inclusion to the CT-scan results (which is the gold standard)
  Diagnostic performance with sensitivity and specificity calculations for the 'curvilinear' probe and the 'phased-array' probe in the detection of an effusion in trauma patients (FAST protocol).

SECONDARY OUTCOMES:
Performance time | During the FAST echography
  The time taken to perform the ultrasound procedure with the phased-array probe and the curvilinear probe in seconds.
Professional experience in FAST echography | After its first inclusion
  The professional experience (which training) of the doctors carrying out this procedure
Previous experience in FAST echography | After its first inclusion
  Previous ultrasound experience (how many years) of doctors performing this procedure
Diagnostic performance according to the area | After the CT-scan results (which is the gold standard)
  Diagnostic performance of the procedure according to the ultrasound area explored (Morisson pouch, Kholer pouch, pelvis, pericardium, lung bases)

CONTACTS AND LOCATIONS:
Overall Officials: Félix AMIOT, MD, Principal Investigator — Hopital Mémorial France Etats-Unis - Urgences/SAMU/SMUR

IPD SHARING:
Plan to Share IPD: No